CLINICAL TRIAL: NCT00052507
Title: A Phase II Study Of PS-341 In Patients With Metastatic Colorectal Cancer
Brief Title: Bortezomib in Treating Patients With Metastatic or Recurrent Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: PMH-PHL-012; CDR0000258488 (Registry Identifier: PDQ (Physician Data Query)); NCI-5890
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
RATIONALE: Bortezomib may interfere with the growth of tumor cells by blocking the enzymes necessary for cancer cell growth.

PURPOSE: Phase II trial to study the effectiveness of bortezomib in treating patients who have metastatic or recurrent colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of bortezomib, in terms of response rate and stable disease rate, in patients with recurrent or metastatic colorectal cancer.
* Determine the toxicity of this drug in these patients.
* Determine the time to progression and response duration in patients treated with this drug.
* Determine whether there is a relationship between levels of transcription factors NF kappa B and HIF-1 alpha and clinical outcome in patients treated with this drug.

OUTLINE: This is an open-label study.

Patients receive bortezomib IV on days 1, 4, 8, and 11. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 21-41 patients will be accrued for this study within 2-4 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the colon or rectum that is incurable with conventional therapy

  * Metastatic or recurrent disease
* At least 1 unidimensionally measurable lesion
* At least 20 mm by conventional techniques or at least 10 mm by spiral CT scan
* Disease must be accessible to biopsy
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1 OR
* Karnofsky 70-100%

Life expectancy

* More than 3 months

Hematopoietic

* Absolute granulocyte count at least 1,500/mm^3
* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.25 times upper limit of normal (ULN)
* AST or ALT no greater than 3 times ULN (less than 5 times ULN if liver metastases present)

Renal

* Creatinine no greater than 1.25 times UNL OR
* Creatinine clearance at least 50 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled concurrent illness
* No ongoing or active infection
* No other active malignancy within the past 3 years except curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix
* No grade 1 or greater peripheral neuropathy due to prior chemotherapy
* No significant traumatic injury within the past 21 days

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No more than 1 line of prior chemotherapy (including any combination of fluorouracil, irinotecan, and/or oxaliplatin) for metastatic disease
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* Prior adjuvant chemotherapy allowed
* No concurrent cytotoxic chemotherapy

Radiotherapy

* More than 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy to measurable target lesion unless disease progression has occurred after radiotherapy
* No concurrent radiotherapy to the sole site of measurable disease

Surgery

* More than 21 days since prior major surgery

Other

* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-01; Primary Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit M. Oza, MD, Study Chair — Princess Margaret Hospital, Canada
Locations (4):
- Canada (4):
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Princess Margaret Hospital at University Health Network, Toronto, Ontario

REFERENCES:
- [Result] Mackay H, Hedley D, Major P, Townsley C, Mackenzie M, Vincent M, Degendorfer P, Tsao MS, Nicklee T, Birle D, Wright J, Siu L, Moore M, Oza A. A phase II trial with pharmacodynamic endpoints of the proteasome inhibitor bortezomib in patients with metastatic colorectal cancer. Clin Cancer Res. 2005 Aug 1;11(15):5526-33. doi: 10.1158/1078-0432.CCR-05-0081. PMID 16061869